CLINICAL TRIAL: NCT00896480
Title: Clinical Activity, Safety and Immunogenic Properties of Cancer Immunotherapeutic GSK2132231A in Patients With Unresectable and Progressive Metastatic Cutaneous Melanoma
Brief Title: Study of GSK2132231A Antigen-Specific Cancer Immunotherapeutic in Patients With Inoperable Metastatic Cutaneous Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111473; 2008-001301-42 (EudraCT Number)
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Results first posted 2019-09-27 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Melanoma
Keywords: ASCI (Antigen-Specific Cancer Immunotherapeutic); MAGE-A3; Malignant melanoma; Cancer immunotherapeutic
MeSH Terms: conditions — Melanoma; Atypical Squamous Cells of the Cervix

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GSK2132231A Group (Experimental): Subjects, male or female, 18 years of age or older, received up to 24 doses of GSK2132231A intramuscularly in 4 cycles. In Cycle 1 (ending Week 13) 6 doses were administered at 2-week intervals; in Cycle 2 (ending Week 32) 6 doses at 3-week intervals; in Cycle 3 (ending Week 54) 4 doses at 6-week intervals and in Cycle 4 4 doses at 12-week intervals, starting 12 weeks after end of Cycle 3, followed by, after an interruption of treatment of 6 months, 4 doses at 24-week intervals.
  Interventions: Biological: Immunotherapeutic GSK2132231A

INTERVENTIONS:
Biological: Immunotherapeutic GSK2132231A — Administration by intramuscular injection
  Other Names: MAGE-A3 ASCI

SUMMARY:
The clinical objective of this clinical trial is to examine the clinical activity in terms of tumor response and time to treatment failure of the immunotherapeutic product GSK2132231A when given to patients with unresectable and progressive metastatic cutaneous melanoma. The safety of the treatment will also be assessed just as its immunogenicity in terms of the humoral and cellular immune response induced by the GSK2132231A immunotherapeutic. Translational research objectives are to assess the effects of the study treatment in terms of various biological variables.

ELIGIBILITY:
Inclusion Criteria:

1. The patient (male or female) has histologically proven, measurable metastatic cutaneous melanoma in one of the following stages according to the American Joint Committee on Cancer classification of 2002:

   * Stage III in transit, or
   * Stage III unresectable, or
   * Stage IV M1a.
2. There has been documented progression of the patient's disease within the 12 weeks before the first administration of study treatment.
3. The patient presents at screening with at least 3 tumor lesions of diameter >= 0.5 mm.
4. Written informed consent has been obtained from the patient before the performance of any protocol-specific procedure.
5. The patient is >= 18 years of age at the time of signature of informed consent.
6. The patient's tumor shows expression of MAGE-A3 gene in at least one of the two tumor biopsies performed at baseline.
7. The patient's ECOG performance status is 0 or 1.
8. The patient has normal organ functions, as assessed by standard laboratory criteria.
9. If the patient is female, she must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to administration of study treatment, have a negative pregnancy test and continue such precautions during the entire study treatment period and for 2 months after completion of the treatment injection series.
10. In the view of the investigator, the patient can and will comply with the requirements of the protocol.

Exclusion Criteria:

1. The patient has at any time received systemic (bio)-chemotherapy
2. The patient is scheduled to receive any anti-cancer specific treatment, including radiotherapy, immunotherapy, chemotherapy and immunomodulating agents.
3. The patient requires concomitant treatment with systemic corticosteroids, or any other immunosuppressive agents.
4. The patient has received any cancer immunotherapeutic containing a MAGE A3 antigen or any cancer immunotherapeutic for his/her metastatic disease.
5. Use of any investigational or non-registered product (drug or vaccine) other than the study treatment within the 30 days preceding the first dose of study treatment, or planned use during the study period.
6. The patient has (or has had) previous or concomitant malignancies at other sites, except effectively treated malignancy that is considered by the investigator highly likely to have been cured.
7. History of allergic disease or reactions likely to be exacerbated by any component of the study investigational product.
8. The patient has an autoimmune disease such as, but not limited to, neuroinflammatory autoimmune diseases, systemic lupus erythematosus, and inflammatory bowel disease
9. The patient has a family history of congenital or hereditary immunodeficiency.
10. The patient is known to be positive for the human immunodeficiency virus (HIV).
11. The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent, or to comply with the study procedures.
12. The patient has concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
13. For female patients: the patient is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-05-19 (Actual); Primary Completion 2014-11-03 (Actual); Study Completion 2014-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Wilrijk
- France (5):
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Reims
  - GSK Investigational Site, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=16043

REFERENCES:
- [Background] Baurain JF, Robert C, Mortier L, Neyns B, Grange F, Lebbe C, Ulloa-Montoya F, De Sousa Alves PM, Gillet M, Louahed J, Jarnjak S, Lehmann FF. Association of homogeneous inflamed gene signature with a better outcome in patients with metastatic melanoma treated with MAGE-A3 immunotherapeutic. ESMO Open. 2018 Jul 25;3(5):e000384. doi: 10.1136/esmoopen-2018-000384. eCollection 2018. PMID 30094070
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- GSK2132231A Group: Subjects, male or female, 18 years of age or older, received up to 24 doses of GSK2132231A intramuscularly in 4 cycles. In Cycle 1 (ending Week 11) 6 doses were administered at 2-week intervals; in Cycle 2 (ending Week 30) 6 doses at 3-week intervals; in Cycle 3 (ending Week 52) 4 doses at 6-week intervals and in Cycle 4 4 doses at 12-week intervals, starting 12 weeks after end of Cycle 3, followed by, after an interruption of treatment of 6 months, 4 doses at 24-week intervals.
Period: Overall Study
Arm/Group | GSK2132231A Group
Started | 24
Completed | 3
Not Completed | 21
Not completed — Disease progression/recurrence | 21

BASELINE CHARACTERISTICS:
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.4 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Objective Tumor Response (OR) to GSK2132231A Study Treatment
Description: OR was defined as the best Overall Response (OR) in a patient. OR = Complete Response (CR) + Partial Response (PR). Responses were categorized as CR, PR, stable disease (SD), SD/PR, progressive disease (PD) and non-evaluable (NE). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by Magnetic-resonance imaging: Complete Response (CR) = disappearance of all target lesions; Partial Response (PR) = ≥30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD) = neither sufficient shrinkage to be PR, not sufficient increase to qualify for Progressive Disease (PD); PD = ≥20% increase in the sum of largest diameter for target lesions. Best objective response = PR or CR. Disease control = CR, or PR, or SD, or SD/PR.
Time Frame: From Pre-treatment (up to 4 weeks before first treatment) to study end (Year 4), each patient being censored out of the analysis at 1st report of disease progression in assessed lesions
Population: The Total Treated population included all patients who have received at least one Dose of the GSK2132231A study treatment
Measure: Count of Participants; unit: Participants
Groups:
- GSK2132231A GS+/+ Group: Subset of subjects from the GSK2132231A Group having a gene signature positive for two biopsies, as assessed at screening.
- GSK2132231A GS+/- Group: Subset of subjects from the GSK2132231A Group having a gene signature positive for only one biopsies, as assessed at screening.
- GSK2132231A GS- Group: Subset of subjects from the GSK2132231A Group having a gene signature negative for both biopsies, as assessed at screening.
Arm/Group | GSK2132231A GS+/+ Group | GSK2132231A GS+/- Group | GSK2132231A GS- Group
Number analyzed (Participants) | 8 | 8 | 8
Participants
  Best response CR | 2 | 0 | 0
  Best response PR | 1 | 1 | 0
  Best response SD | 0 | 1 | 1
  Best response SD/PR | 1 | 0 | 0
  Best response PD | 4 | 6 | 7
  Best response NE | 0 | 0 | 0
  Best objective response Yes | 3 | 1 | 0
  Best objective response No | 5 | 7 | 8
  Disease Control Yes | 4 | 2 | 1
  Disease Control No | 4 | 6 | 7

2. Primary Outcome: Number of Patients With Mixed Response (MR) to GSK2132231A
Description: Assessment was done based on a set of measurable lesions (MLs) identified at baseline as target lesions (TLs) and non-TLs (NTL) followed up until disease progression. MLs assessed for matching below MR definitions. If evaluability per RECIST: a) MR Type 1= at least (a.l.) 30% decrease in LD in a.l. one TL measured at baseline. Such response occurring in SD/PD status of LD of TL and without appearance of one or more new lesions (= SD/PD with TL regression); b) MR Type 2: appearance of one or more new lesions occurring in SD/PR status of LD of TL (= SD/PR with new lesion). If non-evaluability per RECIST (due to LD<20mm): a) MR Type 1 = a clear decrease in diameters occurring in a.l. one TL measured at baseline. Such response occurring in SD/PD status of LD of (baseline) TL and without appearance of one or more new lesions (= SD/PD with TL regression); b) MR Type 2 = appearance of one or more new lesions occurring in SD/PR status of LD of TL (= SD/PR with new lesion).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A GS+/+ Group | GSK2132231A GS+/- Group | GSK2132231A GS- Group
Number analyzed (Participants) | 8 | 8 | 8
Participants
  Best response CR | 2 | 0 | 0
  Best response PR | 1 | 1 | 0
  Best response MR (SD/PR) | 1 | 1 | 0
  Best response MR (SD/PD) | 2 | 0 | 1
  Best response SD | 0 | 0 | 1
  Best response SD/PD | 0 | 0 | 0
  Best response PD (SPD) | 1 | 1 | 2
  Best response PD (SPD/MR) | 1 | 5 | 4
  Best response NE | 0 | 0 | 0

3. Primary Outcome: Time to Treatment Failure (TTF), by Gene Signature
Description: TTF was defined as withdrawal from treatment with the GSK2132231A study product due to disease progression or death. TTF analysis was performed using the non-parametric Kaplan-Meier method.
Time Frame: From Pre-treatment (up to 4 weeks before first treatment) to study end (Year 4), each patient being censored out of the analysis at 1st report of disease progression or death
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | GSK2132231A GS+/+ Group | GSK2132231A GS+/- Group | GSK2132231A GS- Group
Number analyzed (Participants) | 8 | 8 | 8
Months | 14.8 [2.3 to NA] — Upper limit not calculated as 1 patient (among 8) still under treatment at the time of the analysis. | 2.3 [0.5 to 15] | 2.4 [0.5 to 4.6]

4. Primary Outcome: Anti-MAGE-A3 Antibody Concentrations
Description: Anti-MAGE-A3 antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in ELISA units per millilitre (EL.U/mL). A seropositive patient was defined as a patient whose anti-MAGE-A3 antibody concentration was greater than or equal to 27 EL.U/mL. D=Day W=Week
Time Frame: From Pre-treatment (up to 4 weeks before first treatment) to Concluding visit (CCL: at Week 196 + 30 to 37 days for patients completing the treatment, 1 month after the last Dose administered for patients withdrawn from study treatment before completion)
Population: The ATP population for Immunogenicity included all eligible patients, who have received at least the first 6 GSK2132231A study treatment doses and have provided a result for Immunogenicity measurement within 2 weeks following Dose 6.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK2132231A GS+/+ Group | GSK2132231A GS+/- Group | GSK2132231A GS- Group
Number analyzed (Participants) | 7 | 5 | 6
EL.U/mL
  Anti-MAGE-A3, PRE | 13.9 [6.2 to 31.4] | 15.3 [4.7 to 49.9] | 13.8 [6.1 to 31.3]
  Anti-MAGE-A3, D2: number analyzed (Participants) | 7 | 4 | 6
  Anti-MAGE-A3, D2 | 13.9 [6.2 to 30.8] | 16.8 [3.2 to 86.8] | 14.2 [5.8 to 34.7]
  Anti-MAGE-A3, D7 | 16.1 [6.9 to 37.4] | 18.7 [5.9 to 59.2] | 15.5 [7.3 to 32.7]
  Anti-MAGE-A3, D15: number analyzed (Participants) | 7 | 5 | 5
  Anti-MAGE-A3, D15 | 48.5 [11.6 to 202.6] | 72 [7.4 to 699.2] | 55.1 [5.9 to 512.2]
  Anti-MAGE-A3, D16: number analyzed (Participants) | 7 | 3 | 5
  Anti-MAGE-A3, D16 | 55.4 [11.8 to 260.6] | 102.4 [0.7 to 15279.4] | 62.2 [5.8 to 662.9]
  Anti-MAGE-A3, W5: number analyzed (Participants) | 7 | 4 | 5
  Anti-MAGE-A3, W5 | 1396.9 [234.5 to 8321.5] | 4120.2 [2093.0 to 8111.0] | 1484.1 [736.8 to 2989.6]
  Anti-MAGE-A3, W11: number analyzed (Participants) | 4 | 4 | 4
  Anti-MAGE-A3, W11 | 4161.6 [1542.3 to 11229.3] | 9775.9 [3065.3 to 31177.1] | 6181.6 [3414.2 to 11191.8]
  Anti-MAGE-A3, W13: number analyzed (Participants) | 7 | 4 | 5
  Anti-MAGE-A3, W13 | 7797.4 [4564.5 to 13320.2] | 13789.3 [7278.1 to 26125.3] | 8046.1 [7249.1 to 8930.8]
  Anti-MAGE-A3, W21: number analyzed (Participants) | 7 | 2 | 1
  Anti-MAGE-A3, W21 | 7400.3 [4304.0 to 12724.1] | 12544.5 [371.2 to 423881.3] | 10790.0 [NA to NA] — Range not available, as there was only one subject included in the analysis at this timepoint.
  Anti-MAGE-A3, W32: number analyzed (Participants) | 7 | 2 | 1
  Anti-MAGE-A3, W32 | 6128.0 [3601.6 to 10426.5] | 8384.1 [459.4 to 153006.6] | 9641.0 [NA to NA] — Range not available, as there was only one subject included in the analysis at this timepoint.
  Anti-MAGE-A3, W54: number analyzed (Participants) | 4 | 1 | 0
  Anti-MAGE-A3, W54 | 6542.6 [4660.3 to 9185.1] | 12357 [NA to NA] — Range not available, as there was only one subject included in the analysis at this timepoint. |
  Anti-MAGE-A3, W76: number analyzed (Participants) | 3 | 0 | 0
  Anti-MAGE-A3, W76 | 3539.3 [2578.1 to 4859.0] |  |
  Anti-MAGE-A3, W78: number analyzed (Participants) | 1 | 1 | 0
  Anti-MAGE-A3, W78 | 3869.0 [NA to NA] — Range not available, as there was only one subject included in the analysis at this timepoint. | 9219 [NA to NA] — Range not available, as there was only one subject included in the analysis at this timepoint. |
  Anti-MAGE-A3, W100: number analyzed (Participants) | 2 | 1 | 0
  Anti-MAGE-A3, W100 | 4260.0 [452.7 to 40086.0] | 9230 [NA to NA] — Range not available, as there was only one subject included in the analysis at this timepoint. |
  Anti-MAGE-A3, W102: number analyzed (Participants) | 2 | 1 | 0
  Anti-MAGE-A3, W102 | 4804.1 [1467.6 to 15725.7] | 12030 [NA to NA] — Range not available, as there was only one subject included in the analysis at this timepoint. |
  Anti-MAGE-A3, W124: number analyzed (Participants) | 1 | 1 | 0
  Anti-MAGE-A3, W124 | 1575.0 [NA to NA] — Range not available, as there was only one subject included in the analysis at this timepoint. | 7466 [NA to NA] — Range not available, as there was only one subject included in the analysis at this timepoint. |
  Anti-MAGE-A3, W126: number analyzed (Participants) | 2 | 1 | 0
  Anti-MAGE-A3, W126 | 3699.8 [2894.3 to 4729.5] | 11889 [NA to NA] — Range not available, as there was only one subject included in the analysis at this timepoint. |
  Anti-MAGE-A3, W148: number analyzed (Participants) | 2 | 1 | 0
  Anti-MAGE-A3, W148 | 1754.4 [351.7 to 8751.9] | 8865 [NA to NA] — Range not available, as there was only one subject included in the analysis at this timepoint. |
  Anti-MAGE-A3, W150: number analyzed (Participants) | 2 | 1 | 0
  Anti-MAGE-A3, W150 | 3077.8 [5.3 to 1801276] | 10663.0 [NA to NA] — Range not available, as there was only one subject included in the analysis at this timepoint. |
  Anti-MAGE-A3, W174: number analyzed (Participants) | 2 | 0 | 0
  Anti-MAGE-A3, W174 | 2248.7 [226.4 to 22332.9] |  |
  Anti-MAGE-A3, CCL: number analyzed (Participants) | 2 | 0 | 3
  Anti-MAGE-A3, CCL | 4057.1 [0.1 to 135760000] |  | 10004.8 [4092.9 to 24455.9]

5. Primary Outcome: Number of Seroconverted Patients for Anti-MAGE-A3
Description: Seroconversion was defined as a concentration of antibodies assessed that was greater than the cut-off value for a patient whose concentration of such antibodies was below the cut-off level before the initiation of treatment. Seroconverted patients were those patients with anti-MAGE-A3 antibody concentrations ≥ 27 EL.U/mL.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A GS+/+ Group | GSK2132231A GS+/- Group | GSK2132231A GS- Group
Number analyzed (Participants) | 7 | 5 | 6
Participants
  Anti-MAGE-A3, PRE | 1 | 1 | 1
  Anti-MAGE-A3, D2: number analyzed (Participants) | 7 | 4 | 6
  Anti-MAGE-A3, D2 | 1 | 1 | 1
  Anti-MAGE-A3, D7 | 1 | 2 | 1
  Anti-MAGE-A3, D15: number analyzed (Participants) | 7 | 5 | 5
  Anti-MAGE-A3, D15 | 3 | 3 | 3
  Anti-MAGE-A3, D16: number analyzed (Participants) | 7 | 3 | 5
  Anti-MAGE-A3, D16 | 3 | 2 | 3
  Anti-MAGE-A3, W5: number analyzed (Participants) | 7 | 4 | 5
  Anti-MAGE-A3, W5 | 7 | 4 | 5
  Anti-MAGE-A3, W11: number analyzed (Participants) | 4 | 4 | 4
  Anti-MAGE-A3, W11 | 4 | 4 | 4
  Anti-MAGE-A3, W13: number analyzed (Participants) | 7 | 4 | 5
  Anti-MAGE-A3, W13 | 7 | 4 | 5
  Anti-MAGE-A3, W21: number analyzed (Participants) | 7 | 2 | 1
  Anti-MAGE-A3, W21 | 7 | 2 | 1
  Anti-MAGE-A3, W32: number analyzed (Participants) | 7 | 2 | 1
  Anti-MAGE-A3, W32 | 7 | 2 | 1
  Anti-MAGE-A3, W54: number analyzed (Participants) | 4 | 1 | 0
  Anti-MAGE-A3, W54 | 4 | 1 | 0
  Anti-MAGE-A3, W76: number analyzed (Participants) | 3 | 0 | 0
  Anti-MAGE-A3, W76 | 3 | 0 | 0
  Anti-MAGE-A3, W78: number analyzed (Participants) | 1 | 1 | 0
  Anti-MAGE-A3, W78 | 1 | 1 | 0
  Anti-MAGE-A3, W100: number analyzed (Participants) | 2 | 1 | 0
  Anti-MAGE-A3, W100 | 2 | 1 | 0
  Anti-MAGE-A3, W102: number analyzed (Participants) | 2 | 1 | 0
  Anti-MAGE-A3, W102 | 2 | 1 | 0
  Anti-MAGE-A3, W124: number analyzed (Participants) | 1 | 1 | 0
  Anti-MAGE-A3, W124 | 1 | 1 | 0
  Anti-MAGE-A3, W126: number analyzed (Participants) | 2 | 1 | 0
  Anti-MAGE-A3, W126 | 2 | 1 | 0
  Anti-MAGE-A3, W148: number analyzed (Participants) | 2 | 1 | 0
  Anti-MAGE-A3, W148 | 2 | 1 | 0
  Anti-MAGE-A3, W150: number analyzed (Participants) | 2 | 1 | 0
  Anti-MAGE-A3, W150 | 2 | 1 | 0
  Anti-MAGE-A3, W174: number analyzed (Participants) | 2 | 0 | 0
  Anti-MAGE-A3, W174 | 2 | 0 | 0
  Anti-MAGE-A3, CCL: number analyzed (Participants) | 2 | 0 | 3
  Anti-MAGE-A3, CCL | 2 | 0 | 3

6. Primary Outcome: Number of Patients With Treatment Response for Anti-MAGE-A3 Antibodies
Description: For initially seronegative patients: post-administration antibody concentration ≥ 27 EL.U/mL For initially seropositive patients: post-administration antibody concentration ≥ 2 fold the pre-vaccination antibody concentration
Time Frame: From Day 2 to Concluding visit (CCL:at Week 196 + 30 to 37 days for patients completing the treatment, 1 month after the last Dose administered for patients withdrawn from study treatment before completion)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A GS+/+ Group | GSK2132231A GS+/- Group | GSK2132231A GS- Group
Number analyzed (Participants) | 7 | 5 | 6
Participants
  Anti-MAGE-A3, D2: number analyzed (Participants) | 7 | 4 | 6
  Anti-MAGE-A3, D2 | 0 | 0 | 0
  Anti-MAGE-A3, D7 | 0 | 1 | 0
  Anti-MAGE-A3, D15: number analyzed (Participants) | 7 | 5 | 5
  Anti-MAGE-A3, D15 | 3 | 3 | 3
  Anti-MAGE-A3, D16: number analyzed (Participants) | 7 | 3 | 5
  Anti-MAGE-A3, D16 | 3 | 2 | 3
  Anti-MAGE-A3, W5: number analyzed (Participants) | 7 | 4 | 5
  Anti-MAGE-A3, W5 | 7 | 4 | 5
  Anti-MAGE-A3, W11: number analyzed (Participants) | 4 | 4 | 4
  Anti-MAGE-A3, W11 | 4 | 4 | 4
  Anti-MAGE-A3, W13: number analyzed (Participants) | 7 | 4 | 5
  Anti-MAGE-A3, W13 | 7 | 4 | 5
  Anti-MAGE-A3, W21: number analyzed (Participants) | 7 | 2 | 1
  Anti-MAGE-A3, W21 | 7 | 2 | 1
  Anti-MAGE-A3, W32: number analyzed (Participants) | 7 | 2 | 1
  Anti-MAGE-A3, W32 | 7 | 2 | 1
  Anti-MAGE-A3, W54: number analyzed (Participants) | 4 | 1 | 0
  Anti-MAGE-A3, W54 | 4 | 1 | 0
  Anti-MAGE-A3, W76: number analyzed (Participants) | 3 | 0 | 0
  Anti-MAGE-A3, W76 | 3 | 0 | 0
  Anti-MAGE-A3, W78: number analyzed (Participants) | 1 | 1 | 0
  Anti-MAGE-A3, W78 | 1 | 1 | 0
  Anti-MAGE-A3, W100: number analyzed (Participants) | 2 | 1 | 0
  Anti-MAGE-A3, W100 | 2 | 1 | 0
  Anti-MAGE-A3, W102: number analyzed (Participants) | 2 | 1 | 0
  Anti-MAGE-A3, W102 | 2 | 1 | 0
  Anti-MAGE-A3, W124: number analyzed (Participants) | 1 | 1 | 0
  Anti-MAGE-A3, W124 | 1 | 1 | 0
  Anti-MAGE-A3, W126: number analyzed (Participants) | 2 | 1 | 0
  Anti-MAGE-A3, W126 | 2 | 1 | 0
  Anti-MAGE-A3, W148: number analyzed (Participants) | 2 | 1 | 0
  Anti-MAGE-A3, W148 | 2 | 1 | 0
  Anti-MAGE-A3, W150: number analyzed (Participants) | 2 | 1 | 0
  Anti-MAGE-A3, W150 | 2 | 1 | 0
  Anti-MAGE-A3, W174: number analyzed (Participants) | 2 | 0 | 0
  Anti-MAGE-A3, W174 | 2 | 0 | 0
  Anti-MAGE-A3, CCL: number analyzed (Participants) | 2 | 0 | 3
  Anti-MAGE-A3, CCL | 2 | 0 | 3

7. Primary Outcome: Geometric Mean Titers of Anti-MAGE-A3 Specific CD4+ and CD8+ T-cells Concentrations After Immunization
Description: This endpoint presents the geometric mean concentration, expressed in titers, of anti-MAGE-A3 specific CD4+ and CD8+ T-cells. These specific T-cells included the cluster of differentiation 4+ (CD4+) and CD8+ T-cells producing cytokines Tumor Necrosis Factor-alpha (TNF-α) and/or Interferon-gamma (INF-γ).
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 18
Titers
  CD4.TNFα (+) + IFNγ (+) PRE: number analyzed (Participants) | 17
  CD4.TNFα (+) + IFNγ (+) PRE | 1.05 [0.98 to 1.11]
  CD8.TNFα (+) + IFNγ (+) PRE | 1.01 [0.99 to 1.03]
  CD4.TNFα (+) + IFNγ (+) W5: number analyzed (Participants) | 17
  CD4.TNFα (+) + IFNγ (+) W5 | 3.36 [2.2 to 5.13]
  CD8.TNFα (+) + IFNγ (+) W5: number analyzed (Participants) | 17
  CD8.TNFα (+) + IFNγ (+) W5 | 1 [1 to 1]
  CD4.TNFα (+) + IFNγ (+) W13: number analyzed (Participants) | 14
  CD4.TNFα (+) + IFNγ (+) W13 | 5.35 [2.42 to 11.79]
  CD8.TNFα (+) + IFNγ (+) W13: number analyzed (Participants) | 15
  CD8.TNFα (+) + IFNγ (+) W13 | 1 [1 to 1]
  CD4.TNFα (+) + IFNγ (+) W32: number analyzed (Participants) | 10
  CD4.TNFα (+) + IFNγ (+) W32 | 5.29 [2.09 to 13.37]
  CD8.TNFα (+) + IFNγ (+) W32: number analyzed (Participants) | 10
  CD8.TNFα (+) + IFNγ (+) W32 | 1.04 [0.99 to 1.09]
  CD4.TNFα (+) + IFNγ (+) W54: number analyzed (Participants) | 5
  CD4.TNFα (+) + IFNγ (+) W54 | 2.83 [1.04 to 7.68]
  CD8.TNFα (+) + IFNγ (+) W54: number analyzed (Participants) | 5
  CD8.TNFα (+) + IFNγ (+) W54 | 1 [1 to 1]
  CD4.TNFα (+) + IFNγ (+) W78: number analyzed (Participants) | 2
  CD4.TNFα (+) + IFNγ (+) W78 | 2.62 [0.07 to 92.58]
  CD8.TNFα (+) + IFNγ (+) W78: number analyzed (Participants) | 2
  CD8.TNFα (+) + IFNγ (+) W78 | 1 [1 to 1]
  CD4.TNFα (+) + IFNγ (+) W102: number analyzed (Participants) | 3
  CD4.TNFα (+) + IFNγ (+) W102 | 2.13 [0.29 to 15.91]
  CD8.TNFα (+) + IFNγ (+) W102: number analyzed (Participants) | 3
  CD8.TNFα (+) + IFNγ (+) W102 | 1.05 [0.86 to 1.28]
  CD4.TNFα (+) + IFNγ (+) CCL: number analyzed (Participants) | 2
  CD4.TNFα (+) + IFNγ (+) CCL | 2.42 [0 to 185163.6]
  CD8.TNFα (+) + IFNγ (+) CCL: number analyzed (Participants) | 2
  CD8.TNFα (+) + IFNγ (+) CCL | 1 [1 to 1]

8. Primary Outcome: Number of Patients With CD4+ and CD8+ T Cell Frequency ≥ 1.24 Cut-off
Description: A patient was considered as a cellular mediated immune (CMI) responder if there was an increased amount of antigen-specific T-cells after immunization as compared to the patient's baseline value. These specific T-cells included the cluster of differentiation 4+ (CD4+) and CD8+ T-cells producing cytokines Tumor Necrosis Factor-alpha (TNF-α) and/or Interferon-gamma (INF-γ).
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 18
Participants
  CD4.TNFα (+) + IFNγ (+) PRE: number analyzed (Participants) | 17
  CD4.TNFα (+) + IFNγ (+) PRE | 1
  CD8.TNFα (+) + IFNγ (+) PRE | 1
  CD4.TNFα (+) + IFNγ (+) W5: number analyzed (Participants) | 17
  CD4.TNFα (+) + IFNγ (+) W5 | 15
  CD8.TNFα (+) + IFNγ (+) W5: number analyzed (Participants) | 17
  CD8.TNFα (+) + IFNγ (+) W5 | 0
  CD4.TNFα (+) + IFNγ (+) W13: number analyzed (Participants) | 14
  CD4.TNFα (+) + IFNγ (+) W13 | 11
  CD8.TNFα (+) + IFNγ (+) W13: number analyzed (Participants) | 15
  CD8.TNFα (+) + IFNγ (+) W13 | 0
  CD4.TNFα (+) + IFNγ (+) W32: number analyzed (Participants) | 10
  CD4.TNFα (+) + IFNγ (+) W32 | 9
  CD8.TNFα (+) + IFNγ (+) W32: number analyzed (Participants) | 10
  CD8.TNFα (+) + IFNγ (+) W32 | 2
  CD4.TNFα (+) + IFNγ (+) W54: number analyzed (Participants) | 5
  CD4.TNFα (+) + IFNγ (+) W54 | 4
  CD8.TNFα (+) + IFNγ (+) W54: number analyzed (Participants) | 5
  CD8.TNFα (+) + IFNγ (+) W54 | 0
  CD4.TNFα (+) + IFNγ (+) W78: number analyzed (Participants) | 2
  CD4.TNFα (+) + IFNγ (+) W78 | 2
  CD8.TNFα (+) + IFNγ (+) W78: number analyzed (Participants) | 2
  CD8.TNFα (+) + IFNγ (+) W78 | 0
  CD4.TNFα (+) + IFNγ (+) W102: number analyzed (Participants) | 3
  CD4.TNFα (+) + IFNγ (+) W102 | 2
  CD8.TNFα (+) + IFNγ (+) W102: number analyzed (Participants) | 3
  CD8.TNFα (+) + IFNγ (+) W102 | 1
  CD4.TNFα (+) + IFNγ (+) CCL: number analyzed (Participants) | 2
  CD4.TNFα (+) + IFNγ (+) CCL | 1
  CD8.TNFα (+) + IFNγ (+) CCL: number analyzed (Participants) | 2
  CD8.TNFα (+) + IFNγ (+) CCL | 0
  CD4.TNFα (+) + IFNγ (+) At any time point: number analyzed (Participants) | 17
  CD4.TNFα (+) + IFNγ (+) At any time point | 15
  CD8.TNFα (+) + IFNγ (+) At any time point: number analyzed (Participants) | 17
  CD8.TNFα (+) + IFNγ (+) At any time point | 3

9. Primary Outcome: Number of Patients With a Cellular Response (Anti-MAGE-A3 Specific CD4+ and CD8+ T-cells Concentrations After Immunization)
Description: as for outcome 8
Time Frame: From Week 5 to Concluding visit (CCL: at Week 196 + 30 to 37 days for patients completing the treatment, 1 month after the last Dose administered for patients withdrawn from study treatment before completion)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 17
Participants
  CD4.TNFα (+) + IFNγ (+) W5: number analyzed (Participants) | 16
  CD4.TNFα (+) + IFNγ (+) W5 | 5
  CD8.TNFα (+) + IFNγ (+) W5 | 0
  CD4.TNFα (+) + IFNγ (+) W13: number analyzed (Participants) | 13
  CD4.TNFα (+) + IFNγ (+) W13 | 8
  CD8.TNFα (+) + IFNγ (+) W13: number analyzed (Participants) | 15
  CD8.TNFα (+) + IFNγ (+) W13 | 0
  CD4.TNFα (+) + IFNγ (+) W32: number analyzed (Participants) | 9
  CD4.TNFα (+) + IFNγ (+) W32 | 4
  CD8.TNFα (+) + IFNγ (+) W32: number analyzed (Participants) | 10
  CD8.TNFα (+) + IFNγ (+) W32 | 0
  CD4.TNFα (+) + IFNγ (+) W54: number analyzed (Participants) | 4
  CD4.TNFα (+) + IFNγ (+) W54 | 2
  CD8.TNFα (+) + IFNγ (+) W54: number analyzed (Participants) | 5
  CD8.TNFα (+) + IFNγ (+) W54 | 0
  CD4.TNFα (+) + IFNγ (+) W78: number analyzed (Participants) | 2
  CD4.TNFα (+) + IFNγ (+) W78 | 0
  CD8.TNFα (+) + IFNγ (+) W78: number analyzed (Participants) | 2
  CD8.TNFα (+) + IFNγ (+) W78 | 0
  CD4.TNFα (+) + IFNγ (+) W102: number analyzed (Participants) | 3
  CD4.TNFα (+) + IFNγ (+) W102 | 1
  CD8.TNFα (+) + IFNγ (+) W102: number analyzed (Participants) | 3
  CD8.TNFα (+) + IFNγ (+) W102 | 0
  CD4.TNFα (+) + IFNγ (+) CCL: number analyzed (Participants) | 2
  CD4.TNFα (+) + IFNγ (+) CCL | 1
  CD8.TNFα (+) + IFNγ (+) CCL: number analyzed (Participants) | 2
  CD8.TNFα (+) + IFNγ (+) CCL | 0
  CD4.TNFα (+) + IFNγ (+) At any time point: number analyzed (Participants) | 16
  CD4.TNFα (+) + IFNγ (+) At any time point | 12
  CD8.TNFα (+) + IFNγ (+) At any time point | 0

10. Primary Outcome: Number of Patients Reported With Antigen Specific Cancer Immunotherapeutics (ASCI)-Related grade3/4 Adverse Events (AEs) According to the Common Terminology Criteria (CTCAE) Version 3.0.
Description: The assessed AEs were ASCI-related grade 3/4 adverse events according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. An unsolicited AE covers any untoward medical occurrence in a clinical investigation patient temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e. lack of efficacy), abuse or misuse. AEs may include pre- or post-treatment events that occur as a result of protocol-mandated procedures (i.e. invasive procedures, modification of patient's previous therapeutic regimen).
Time Frame: Within the 31-day (Days 0-30) post-administration periods
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  Any event, Grade 3 | 0
  Any event, Grade 4 | 0

11. Primary Outcome: Number of Patients Reported With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a patient, is a Grade 4 AE according to the CTCAE, version3.0. Events which were part of the natural course of the disease under study were captured as part of the clinical activity outcome variables in this study; therefore did not need to be reported as SAEs. Progression/recurrence of the tumor was recorded as part of the clinical assessment data collection, and deaths due to progressive disease was recorded on a specific form, but not as an SAE. However, if the investigator considered that there was a causal relationship between treatment or protocol design/procedures and the disease progression/recurrence, then the event was reported as an SAE. Any new primary cancer (non-related to the cancer under study) was reported as an SAE.
Time Frame: During the entire study period (from Day 0 to CCL: at Week 196 + 30 to 37 days for patients completing the treatment, 1 month after the last Dose administered for patients withdrawn from study treatment before completion
Population: The Total Treated population included all patients who have received at least one Dose of the GSK2132231A ASCI study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants | 2

12. Primary Outcome: Number of Patients With Abnormal Alanine Aminotransferase (ALT) Values by Maximum Grade
Description: The status of each patient was collected and graded according to the Common Terminology Criteria Adverse Event (CTCAE v.03) terminology. Gradings were: G0 (normal value), G1 (Mild abnormality), G2 (Moderate abnormality), G3 (Severe abnormality), G4 (Life-threatening/Disabling abnormality), Unknown abnormality (UNK).
  The post-treatment values, at Study End (SE) were presented versus baseline values, at Screening (SCR). [e.g. ALT - SCR G0; SE G3 = ALT with no abnormality/normal value at screening and with Severe abnormality at study end].
Time Frame: From Screening and up to Week 11 (Cycle 1), Week 30 (Cycle 2), Week 52 (Cycle 3), and Study End at Year 4 (Cycle 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  ALT - SCR G0; SE G0 | 20
  ALT - SCR G0; SE G1 | 3
  ALT - SCR G0; SE G2 | 0
  ALT - SCR G0; SE G3 | 1
  ALT - SCR G0; SE G4 | 0
  ALT - SCR G0; SE UNK | 0

13. Primary Outcome: Number of Patients With Abnormal Aspartate Aminotransferase (AST) Values by Maximum Grade
Description: The status of each patient was collected and graded according to the Common Terminology Criteria Adverse Event (CTCAE v.03) terminology. Gradings were: G0 (normal value), G1 (Mild abnormality), G2 (Moderate abnormality), G3 (Severe abnormality), G4 (Life-threatening/Disabling abnormality), Unknown abnormality (UNK).
  The post-treatment values, at Study End (SE) were presented versus baseline values, at Screening (SCR). [e.g. AST - SCR G0; SE G3 = AST with no abnormality/normal value at screening and with Severe abnormality at study end].
Time Frame: From Screening and up to Week 11 (Cycle 1), Week 30 (Cycle 2), Week 52 (Cycle 3), and Study End at Year 4 (Cycle 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  AST - SCR G0; SE G0 | 19
  AST - SCR G0; SE G1 | 5
  AST - SCR G0; SE G2 | 0
  AST - SCR G0; SE G3 | 0
  AST - SCR G0; SE G4 | 0
  AST - SCR G0; SE UNK | 0

14. Primary Outcome: Number of Patients With Abnormal Alkaline Phosphatase (ALK) Values by Maximum Grade
Description: The status of each patient was collected and graded according to the Common Terminology Criteria Adverse Event (CTCAE v.03) terminology. Gradings were: G0 (normal value), G1 (Mild abnormality), G2 (Moderate abnormality), G3 (Severe abnormality), G4 (Life-threatening/Disabling abnormality), Unknown abnormality (UNK).
  The post-treatment values, at Study End (SE) were presented versus baseline values, at Screening (SCR). [e.g. ALK - SCR G0; SE G3 = ALK with no abnormality/normal value at screening and with Severe abnormality at study end].
Time Frame: From Screening and up to Week 11 (Cycle 1), Week 30 (Cycle 2), Week 52 (Cycle 3), and Study End at Year 4 (Cycle 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  ALK - SCR UNK; SE G0 | 0
  ALK - SCR UNK; SE G1 | 0
  ALK - SCR UNK; SE G2 | 0
  ALK - SCR UNK; SE G3 | 0
  ALK - SCR UNK; SE G4 | 0
  ALK - SCR UNK; SE UNK | 1
  ALK - SCR G0; SE G0 | 17
  ALK - SCR G0; SE G1 | 6
  ALK - SCR G0; SE G2 | 0
  ALK - SCR G0; SE G3 | 0
  ALK - SCR G0; SE G4 | 0
  ALK - SCR G0; SE UNK | 0

15. Primary Outcome: Number of Patients With Abnormal Bilirubine (BIL) Values by Maximum Grade
Description: The status of each patient was collected and graded according to the Common Terminology Criteria Adverse Event (CTCAE v.03) terminology. Gradings were: G0 (normal value), G1 (Mild abnormality), G2 (Moderate abnormality), G3 (Severe abnormality), G4 (Life-threatening/Disabling abnormality), Unknown abnormality (UNK).
  The post-treatment values, at Study End (SE) were presented versus baseline values, at Screening (SCR). [e.g. BIL - SCR G0; SE G3 = BIL with no abnormality/normal value at screening and with Severe abnormality at study end].
Time Frame: From Screening and up to Week 11 (Cycle 1), Week 30 (Cycle 2), Week 52 (Cycle 3), and Study End at Year 4 (Cycle 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  BIL - SCR G0; SE G0 | 24
  BIL - SCR G0; SE G1 | 0
  BIL - SCR G0; SE G2 | 0
  BIL - SCR G0; SE G3 | 0
  BIL - SCR G0; SE G4 | 0
  BIL - SCR G0; SE UNK | 0

16. Primary Outcome: Number of Patients With Abnormal Creatinine (CREA) Values by Maximum Grade
Description: The status of each patient was collected and graded according to the Common Terminology Criteria Adverse Event (CTCAE v.03) terminology. Gradings were: G0 (normal value), G1 (Mild abnormality), G2 (Moderate abnormality), G3 (Severe abnormality), G4 (Life-threatening/Disabling abnormality), Unknown abnormality (UNK).
  The post-treatment values, at Study End (SE) were presented versus baseline values, at Screening (SCR). [e.g. CREA - SCR G0; SE G3 = CREA with no abnormality/normal value at screening and with Severe abnormality at study end].
Time Frame: From Screening and up to Week 11 (Cycle 1), Week 30 (Cycle 2), Week 52 (Cycle 3), and Study End at Year 4 (Cycle 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  CREA - SCR G0; SE G0 | 20
  CREA - SCR G0; SE G1 | 2
  CREA - SCR G0; SE G2 | 0
  CREA - SCR G0; SE G3 | 0
  CREA - SCR G0; SE G4 | 0
  CREA - SCR G0; SE UNK | 1
  CREA - SCR G1; SE G0 | 0
  CREA - SCR G1; SE G1 | 0
  CREA - SCR G1; SE G2 | 1
  CREA - SCR G1; SE G3 | 0
  CREA - SCR G1; SE G4 | 0
  CREA - SCR G1; SE UNK | 0

17. Primary Outcome: Number of Patients With Abnormal Gamma-glutamyl Transpeptidase (GGT) Values by Maximum Grade
Description: The status of each patient was collected and graded according to the Common Terminology Criteria Adverse Event (CTCAE v.03) terminology. Gradings were: G0 (normal value), G1 (Mild abnormality), G2 (Moderate abnormality), G3 (Severe abnormality), G4 (Life-threatening/Disabling abnormality), Unknown abnormality (UNK).
  The post-treatment values, at Study End (SE) were presented versus baseline values, at Screening (SCR). [e.g. GGT - SCR G0; SE G3 = GGT with no abnormality/normal value at screening and with Severe abnormality at study end].
Time Frame: From Screening and up to Week 11 (Cycle 1), Week 30 (Cycle 2), Week 52 (Cycle 3), and Study End at Year 4 (Cycle 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  GGT - SCR UNK; SE G0 | 0
  GGT - SCR UNK; SE G1 | 1
  GGT - SCR UNK; SE G2 | 0
  GGT - SCR UNK; SE G3 | 0
  GGT - SCR UNK; SE G4 | 0
  GGT - SCR UNK; SE UNK | 0
  GGT - SCR G0; SE G0 | 17
  GGT - SCR G0; SE G1 | 2
  GGT - SCR G0; SE G2 | 1
  GGT - SCR G0; SE G3 | 0
  GGT - SCR G0; SE G4 | 0
  GGT - SCR G0; SE UNK | 0
  GGT - SCR G1; SE G0 | 0
  GGT - SCR G1; SE G1 | 2
  GGT - SCR G1; SE G2 | 0
  GGT - SCR G1; SE G3 | 1
  GGT - SCR G1; SE G4 | 0
  GGT - SCR G1; SE UNK | 0

18. Primary Outcome: Number of Patients With Abnormal Hemoglobin (HGB) Values by Maximum Grade
Description: The status of each patient was collected and graded according to the Common Terminology Criteria Adverse Event (CTCAE v.03) terminology. Gradings were: G0 (normal value), G1 (Mild abnormality), G2 (Moderate abnormality), G3 (Severe abnormality), G4 (Life-threatening/Disabling abnormality), Unknown abnormality (UNK).
  The post-treatment values, at Study End (SE) were presented versus baseline values, at Screening (SCR). [e.g. HGB - SCR G0; SE G3 = HGB with no abnormality/normal value at screening and with Severe abnormality at study end].
Time Frame: From Screening and up to Week 11 (Cycle 1), Week 30 (Cycle 2), Week 52 (Cycle 3), and Study End at Year 4 (Cycle 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  HGB - SCR G0; SE G0 | 14
  HGB - SCR G0; SE G1 | 9
  HGB - SCR G0; SE G2 | 0
  HGB - SCR G0; SE G3 | 0
  HGB - SCR G0; SE G4 | 0
  HGB - SCR G0; SE UNK | 0
  HGB - SCR G1; SE G0 | 0
  HGB - SCR G1; SE G1 | 1
  HGB - SCR G1; SE G2 | 0
  HGB - SCR G1; SE G3 | 0
  HGB - SCR G1; SE G4 | 0
  HGB - SCR G1; SE UNK | 0

19. Primary Outcome: Number of Patients With Abnormal Hypercalcemia (HCA) Values by Maximum Grade
Description: The status of each patient was collected and graded according to the Common Terminology Criteria Adverse Event (CTCAE v.03) terminology. Gradings were: G0 (normal value), G1 (Mild abnormality), G2 (Moderate abnormality), G3 (Severe abnormality), G4 (Life-threatening/Disabling abnormality), Unknown abnormality (UNK).
  The post-treatment values, at Study End (SE) were presented versus baseline values, at Screening (SCR). [e.g. HCA - SCR G0; SE G3 = HCA with no abnormality/normal value at screening and with Severe abnormality at study end].
Time Frame: From Screening and up to Week 11 (Cycle 1), Week 30 (Cycle 2), Week 52 (Cycle 3), and Study End at Year 4 (Cycle 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  HCA - SCR UNK; SE G0 | 3
  HCA - SCR UNK; SE G1 | 0
  HCA - SCR UNK; SE G2 | 0
  HCA - SCR UNK; SE G3 | 0
  HCA - SCR UNK; SE G4 | 0
  HCA - SCR UNK; SE UNK | 0
  HCA - SCR G0; SE G0 | 15
  HCA - SCR G0; SE G1 | 3
  HCA - SCR G0; SE G2 | 0
  HCA - SCR G0; SE G3 | 0
  HCA - SCR G0; SE G4 | 0
  HCA - SCR G0; SE UNK | 0
  HCA - SCR G1; SE G0 | 1
  HCA - SCR G1; SE G1 | 2
  HCA - SCR G1; SE G2 | 0
  HCA - SCR G1; SE G3 | 0
  HCA - SCR G1; SE G4 | 0
  HCA - SCR G1; SE UNK | 0

20. Primary Outcome: Number of Patients With Abnormal Hyperkalemia (HKA) Values by Maximum Grade
Description: The status of each patient was collected and graded according to the Common Terminology Criteria Adverse Event (CTCAE v.03) terminology. Gradings were: G0 (normal value), G1 (Mild abnormality), G2 (Moderate abnormality), G3 (Severe abnormality), G4 (Life-threatening/Disabling abnormality), Unknown abnormality (UNK).
  The post-treatment values, at Study End (SE) were presented versus baseline values, at Screening (SCR). [e.g. HKA - SCR G0; SE G3 = HKA with no abnormality/normal value at screening and with Severe abnormality at study end].
Time Frame: From Screening and up to Week 11 (Cycle 1), Week 30 (Cycle 2), Week 52 (Cycle 3), and Study End at Year 4 (Cycle 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  HKA - SCR UNK; SE G0 | 2
  HKA - SCR UNK; SE G1 | 0
  HKA - SCR UNK; SE G2 | 0
  HKA - SCR UNK; SE G3 | 0
  HKA - SCR UNK; SE G4 | 0
  HKA - SCR UNK; SE UNK | 0
  HKA - SCR G0; SE G0 | 17
  HKA - SCR G0; SE G1 | 3
  HKA - SCR G0; SE G2 | 1
  HKA - SCR G0; SE G3 | 0
  HKA - SCR G0; SE G4 | 0
  HKA - SCR G0; SE UNK | 0
  HKA - SCR G1; SE G0 | 0
  HKA - SCR G1; SE G1 | 0
  HKA - SCR G1; SE G2 | 1
  HKA - SCR G1; SE G3 | 0
  HKA - SCR G1; SE G4 | 0
  HKA - SCR G1; SE UNK | 0

21. Primary Outcome: Number of Patients With Abnormal Hypernatremia (HNA) Values by Maximum Grade
Description: The status of each patient was collected and graded according to the Common Terminology Criteria Adverse Event (CTCAE v.03) terminology. Gradings were: G0 (normal value), G1 (Mild abnormality), G2 (Moderate abnormality), G3 (Severe abnormality), G4 (Life-threatening/Disabling abnormality), Unknown abnormality (UNK).
  The post-treatment values, at Study End (SE) were presented versus baseline values, at Screening (SCR). [e.g. HNA - SCR G0; SE G3 = HNA with no abnormality/normal value at screening and with Severe abnormality at study end].
Time Frame: From Screening and up to Week 11 (Cycle 1), Week 30 (Cycle 2), Week 52 (Cycle 3), and Study End at Year 4 (Cycle 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  HNA - SCR UNK; SE G0 | 2
  HNA - SCR UNK; SE G1 | 0
  HNA - SCR UNK; SE G2 | 0
  HNA - SCR UNK; SE G3 | 0
  HNA - SCR UNK; SE G4 | 0
  HNA - SCR UNK; SE UNK | 0
  HNA - SCR G0; SE G0 | 19
  HNA - SCR G0; SE G1 | 3
  HNA - SCR G0; SE G2 | 0
  HNA - SCR G0; SE G3 | 0
  HNA - SCR G0; SE G4 | 0
  HNA - SCR G0; SE UNK | 0

22. Primary Outcome: Number of Patients With Abnormal Hypoalbuminemia (hAL) Values by Maximum Grade
Description: The status of each patient was collected and graded according to the Common Terminology Criteria Adverse Event (CTCAE v.03) terminology. Gradings were: G0 (normal value), G1 (Mild abnormality), G2 (Moderate abnormality), G3 (Severe abnormality), G4 (Life-threatening/Disabling abnormality), Unknown abnormality (UNK).
  The post-treatment values, at Study End (SE) were presented versus baseline values, at Screening (SCR). [e.g. hAL - SCR G0; SE G3 = hAL with no abnormality/normal value at screening and with Severe abnormality at study end].
Time Frame: From Screening and up to Week 11 (Cycle 1), Week 30 (Cycle 2), Week 52 (Cycle 3), and Study End at Year 4 (Cycle 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  hAL - SCR UNK; SE G0 | 1
  hAL - SCR UNK; SE G1 | 1
  hAL - SCR UNK; SE G2 | 0
  hAL - SCR UNK; SE G3 | 0
  hAL - SCR UNK; SE G4 | 0
  hAL - SCR UNK; SE UNK | 0
  hAL - SCR G0; SE G0 | 21
  hAL - SCR G0; SE G1 | 0
  hAL - SCR G0; SE G2 | 0
  hAL - SCR G0; SE G3 | 0
  hAL - SCR G0; SE G4 | 0
  hAL - SCR G0; SE UNK | 1

23. Primary Outcome: Number of Patients With Abnormal Hypocalcemia (hCA) Values by Maximum Grade
Description: as for outcome 19
Time Frame: From Screening and up to Week 11 (Cycle 1), Week 30 (Cycle 2), Week 52 (Cycle 3), and Study End at Year 4 (Cycle 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  hCA - SCR UNK; SE G0 | 3
  hCA - SCR UNK; SE G1 | 0
  hCA - SCR UNK; SE G2 | 0
  hCA - SCR UNK; SE G3 | 0
  hCA - SCR UNK; SE G4 | 0
  hCA - SCR UNK; SE UNK | 0
  hCA - SCR G0; SE G0 | 18
  hCA - SCR G0; SE G1 | 2
  hCA - SCR G0; SE G2 | 0
  hCA - SCR G0; SE G3 | 0
  hCA - SCR G0; SE G4 | 0
  hCA - SCR G0; SE UNK | 0
  hCA - SCR G1; SE G0 | 0
  hCA - SCR G1; SE G1 | 1
  hCA - SCR G1; SE G2 | 0
  hCA - SCR G1; SE G3 | 0
  hCA - SCR G1; SE G4 | 0
  hCA - SCR G1; SE UNK | 0

24. Primary Outcome: Number of Patients With Abnormal Hypokalemia (hKA) Values by Maximum Grade
Description: as for outcome 20
Time Frame: From Screening and up to Week 11 (Cycle 1), Week 30 (Cycle 2), Week 52 (Cycle 3), and Study End at Year 4 (Cycle 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  hKA - SCR UNK; SE G0 | 2
  hKA - SCR UNK; SE G1 | 0
  hKA - SCR UNK; SE G2 | 0
  hKA - SCR UNK; SE G3 | 0
  hKA - SCR UNK; SE G4 | 0
  hKA - SCR UNK; SE UNK | 0
  hKA - SCR G0; SE G0 | 19
  hKA - SCR G0; SE G1 | 3
  hKA - SCR G0; SE G2 | 0
  hKA - SCR G0; SE G3 | 0
  hKA - SCR G0; SE G4 | 0
  hKA - SCR G0; SE UNK | 0

25. Primary Outcome: Number of Patients With Abnormal Hyponatremia (hNA) Values by Maximum Grade
Description: as for outcome 21
Time Frame: From Screening and up to Week 11 (Cycle 1), Week 30 (Cycle 2), Week 52 (Cycle 3), and Study End at Year 4 (Cycle 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  hNA - SCR UNK; SE G0 | 2
  hNA - SCR UNK; SE G1 | 0
  hNA - SCR UNK; SE G2 | 0
  hNA - SCR UNK; SE G3 | 0
  hNA - SCR UNK; SE G4 | 0
  hNA - SCR UNK; SE UNK | 0
  hNA - SCR G0; SE G0 | 18
  hNA - SCR G0; SE G1 | 4
  hNA - SCR G0; SE G2 | 0
  hNA - SCR G0; SE G3 | 0
  hNA - SCR G0; SE G4 | 0
  hNA - SCR G0; SE UNK | 0

26. Primary Outcome: Number of Patients With Abnormal Leukocytes (LEU) Values by Maximum Grade
Description: The status of each patient was collected and graded according to the Common Terminology Criteria Adverse Event (CTCAE v.03) terminology. Gradings were: G0 (normal value), G1 (Mild abnormality), G2 (Moderate abnormality), G3 (Severe abnormality), G4 (Life-threatening/Disabling abnormality), Unknown abnormality (UNK).
  The post-treatment values, at Study End (SE) were presented versus baseline values, at Screening (SCR). [e.g. LEU - SCR G0; SE G3 = LEU with no abnormality/normal value at screening and with Severe abnormality at study end].
Time Frame: From Screening and up to Week 11 (Cycle 1), Week 30 (Cycle 2), Week 52 (Cycle 3), and Study End at Year 4 (Cycle 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  LEU - SCR G0; SE G0 | 21
  LEU - SCR G0; SE G1 | 2
  LEU - SCR G0; SE G2 | 0
  LEU - SCR G0; SE G3 | 0
  LEU - SCR G0; SE G4 | 0
  LEU - SCR G0; SE UNK | 0
  LEU - SCR G1; SE G0 | 1
  LEU - SCR G1; SE G1 | 0
  LEU - SCR G1; SE G2 | 0
  LEU - SCR G1; SE G3 | 0
  LEU - SCR G1; SE G4 | 0
  LEU - SCR G1; SE UNK | 0

27. Primary Outcome: Number of Patients With Abnormal Lymphopenia (LYM) Values by Maximum Grade
Description: The status of each patient was collected and graded according to the Common Terminology Criteria Adverse Event (CTCAE v.03) terminology. Gradings were: G0 (normal value), G1 (Mild abnormality), G2 (Moderate abnormality), G3 (Severe abnormality), G4 (Life-threatening/Disabling abnormality), Unknown abnormality (UNK).
  The post-treatment values, at Study End (SE) were presented versus baseline values, at Screening (SCR). [e.g. LYM - SCR G0; SE G3 = LYM with no abnormality/normal value at screening and with Severe abnormality at study end].
Time Frame: From Screening and up to Week 11 (Cycle 1), Week 30 (Cycle 2), Week 52 (Cycle 3), and Study End at Year 4 (Cycle 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  LYM - SCR G0; SE G0 | 17
  LYM - SCR G0; SE G1 | 0
  LYM - SCR G0; SE G2 | 3
  LYM - SCR G0; SE G3 | 0
  LYM - SCR G0; SE G4 | 0
  LYM - SCR G0; SE UNK | 0
  LYM - SCR G1; SE G0 | 1
  LYM - SCR G1; SE G1 | 3
  LYM - SCR G1; SE G2 | 0
  LYM - SCR G1; SE G3 | 0
  LYM - SCR G1; SE G4 | 0
  LYM - SCR G1; SE UNK | 0

28. Primary Outcome: Number of Patients With Abnormal Neutrophils (NEU) Values by Maximum Grade
Description: The status of each patient was collected and graded according to the Common Terminology Criteria Adverse Event (CTCAE v.03) terminology. Gradings were: G0 (normal value), G1 (Mild abnormality), G2 (Moderate abnormality), G3 (Severe abnormality), G4 (Life-threatening/Disabling abnormality), Unknown abnormality (UNK).
  The post-treatment values, at Study End (SE) were presented versus baseline values, at Screening (SCR). [e.g. NEU - SCR G0; SE G3 = NEU with no abnormality/normal value at screening and with Severe abnormality at study end].
Time Frame: From Screening and up to Week 11 (Cycle 1), Week 30 (Cycle 2), Week 52 (Cycle 3), and Study End at Year 4 (Cycle 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  NEU - SCR G0; SE G0 | 21
  NEU - SCR G0; SE G1 | 2
  NEU - SCR G0; SE G2 | 1
  NEU - SCR G0; SE G3 | 0
  NEU - SCR G0; SE G4 | 0
  NEU - SCR G0; SE UNK | 0

29. Primary Outcome: Number of Patients With Abnormal Platelets (PLT) Values by Maximum Grade
Description: The status of each patient was collected and graded according to the Common Terminology Criteria Adverse Event (CTCAE v.03) terminology. Gradings were: G0 (normal value), G1 (Mild abnormality), G2 (Moderate abnormality), G3 (Severe abnormality), G4 (Life-threatening/Disabling abnormality), Unknown abnormality (UNK).
  The post-treatment values, at Study End (SE) were presented versus baseline values, at Screening (SCR). [e.g. PLT - SCR G0; SE G3 = PLT with no abnormality/normal value at screening and with Severe abnormality at study end].
Time Frame: From Screening and up to Week 11 (Cycle 1), Week 30 (Cycle 2), Week 52 (Cycle 3), and Study End at Year 4 (Cycle 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  PLT - SCR G0; SE G0 | 24
  PLT - SCR G0; SE G1 | 0
  PLT - SCR G0; SE G2 | 0
  PLT - SCR G0; SE G3 | 0
  PLT - SCR G0; SE G4 | 0
  PLT - SCR G0; SE UNK | 0

30. Primary Outcome: Number of Patients With Any Adverse Events (AEs) and With AEs by Maximum Grade
Description: An AE was any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs reported are here below tabulated irrespective of grade (any), as well as graded by maximum grade reported according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. Maximum grade reported and tabulated were Grade 1 (G1) - Mild AE, G2 - Moderate AE, G3 - Severe AE, G4 - Life threatening/Disabling AE and G5 - Death related to AE.
Time Frame: Within the 31-day (Day 0-30) follow-up period post treatment administration.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  Patients with any AEs | 24
  Patients with G1 AEs | 6
  Patients with G2 AEs | 15
  Patients with G3 AEs | 3
  Patients with G4 AEs | 0
  Patients with G5 AEs | 0

31. Primary Outcome: Number of Patients With Any AE(s) and With AEs by Maximum Grade, Related to Treatment Administration
Description: as for outcome 30
Time Frame: Within the 31-day (Day 0-30) follow-up period post treatment administration.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  Patients with any related AEs | 23
  Patients with G1 related AEs | 11
  Patients with G2 related AEs | 12
  Patients with G3 related AEs | 0
  Patients with G4 related AEs | 0
  Patients with G5 related AEs | 0

32. Primary Outcome: Number of Patients With Any Serious Adverse Events (SAEs) and With SAEs by Maximum Grade
Description: SAEs include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a patient. Events which were part of the natural course of the disease under study were captured as part of the clinical activity outcome variables in this study; therefore did not need to be reported as SAEs. Progression/recurrence of the tumor was recorded as part of the clinical assessment data collection, and deaths due to progressive disease was recorded on a specific form, but not as an SAE. SAEs reported are here below tabulated irrespective of grade (any), as well as graded by maximum grade reported according to the CTC Adverse event terminology, version 3.0. Maximum grade reported and tabulated were Grade 1 (G1) - Mild SAE, G2 - Moderate SAE, G3 - Severe SAE, G4 - Life threatening/Disabling SAE and G5 - Death related to SAE.
Time Frame: Within the 31-day (Day 0-30) follow-up period post treatment administration.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  Patients with any SAEs | 2
  Patients with G1 SAEs | 0
  Patients with G2 SAEs | 1
  Patients with G3 SAEs | 1
  Patients with G4 SAEs | 0
  Patients with G5 SAEs | 0

33. Primary Outcome: Number of Patients With Any Serious Adverse Events (SAEs) and With SAEs by Maximum Grade, Related to Treatment Administration
Description: as for outcome 32
Time Frame: Within the 31-day (Day 0-30) follow-up period post treatment administration.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A Group
Number analyzed (Participants) | 24
Participants
  Patients with any related SAEs | 0
  Patients with G1 related SAEs | 0
  Patients with G2 related SAEs | 0
  Patients with G3 related SAEs | 0
  Patients with G4 related SAEs | 0
  Patients with G5 related SAEs | 0

ADVERSE EVENTS:
Time Frame: Unsolicited AEs during the 31-day post-vaccination (Days 0-30), SAEs during the entire study period (Day 0 - Year 4).
Groups:
- GSK2132231A Group: Patients planned to receive intramuscularly up to 24 doses of GSK2132231A (the study product), in 4 cycles.
Arm/Group | GSK2132231A Group
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 2/24
Other Adverse Events (participants affected / at risk) | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2132231A Group (N=24)
Cardiac disorder (Cardiac disorders) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2132231A Group (N=24)
Administration site pain (General disorders) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Asthenia (General disorders) | 9 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Chills (General disorders) | 4 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Discomfort (General disorders) | 3 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Fatigue (General disorders) | 7 (13)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 7 (31)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Influenza like illness (General disorders) | 7 (40)
Injection site erythema (General disorders) | 4 (7)
Injection site induration (General disorders) | 2 (7)
Injection site pain (General disorders) | 12 (40)
Injection site reaction (General disorders) | 12 (50)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (18)
Nausea (Gastrointestinal disorders) | 7 (17)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (7)
Pyrexia (General disorders) | 10 (31)
Skin infection (Infections and infestations) | 2 (2)
Ulcer (General disorders) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.